CLINICAL TRIAL: NCT05669755
Title: The Cardiovascular Safety and Efficacy of Cagrilintide 2.4 mg s.c. in Combination With Semaglutide 2.4 mg s.c. (CagriSema 2.4 mg/2.4 mg s.c.) Once-weekly in Participants With Established Cardiovascular Disease
Brief Title: REDEFINE 3: A Research Study to See the Effects of CagriSema in People Living With Diseases in the Heart and Blood Vessels
Acronym: REDEFINE 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4942; U1111-1270-0943 (Other: World Health Organization (WHO)); 2021-005855-35 (EudraCT Number); jRCT2031220672 (Registry Identifier: jrct (Japan))
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Participants will receive cagrilintide and semaglutide subcutaneously (s.c.) once-weekly after a dose escalation period of 16 weeks during the maintenance period of 219 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive placebo matched to cagrilintide and placebo matched to semaglutide s.c. once weekly for 235 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive cagrilintide s.c. once-weekly after a dose escalation period of 16 weeks for 219 weeks.
  Arms: CagriSema
Drug: Semaglutide — Participants will receive semaglutide s.c. once-weekly after a dose escalation period of 16 weeks for 219 weeks.
  Arms: CagriSema
Drug: Placebo — Participants will receive placebo matched to cagrilintide and placebo matched to semaglutide subcutaneously.
  Arms: Placebo

SUMMARY:
This study will look at the effects of CagriSema on cardiovascular events (for example heart attack and stroke) in people living with cardiovascular disease. Participants will either get CagriSema or a dummy medicine (also called "placebo") which has no effect on the body. Which treatment participants will get will be decided by chance. Participant's chance of getting CagriSema or placebo is the same. Participants will inject the study medicine once a week. The study medicine will be injected briefly with a thin needle, typically in the stomach, thighs or upper arms. The study will last for up to 4.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age above or equal to 55 years at the time of signing informed consent
* Body mass index (BMI) greater than or equal to (>=) 25.0 kilograms per meter square (kg/m^2)
* Established CVD as evidenced by at least one of the following:

  1. Prior myocardial infarction
  2. Prior stroke (ischemic or haemorrhagic stroke)
  3. Symptomatic peripheral arterial disease (PAD) defined as at least one of the following:

     1. Intermittent claudication with an ankle-brachial index (ABI) less than (<) 0.85 at rest
     2. Intermittent claudication with a >= 50% stenosis in a lower extremity peripheral artery documented by X-ray angiography, magnetic resonance (MR) angiography, computed tomography (CT) angiography or Doppler ultrasound
     3. Prior revascularization procedure of a lower extremity peripheral artery
     4. Lower extremity amputation at or above ankle due to atherosclerotic disease (excluding e.g., trauma or osteomyelitis)

For participants with T2D at screening the following inclusion criteria also apply:

* Diagnosed with type 2 diabetes mellitus (T2D) >= 180 days before screening
* HbA1c 6.5%-10% (47-86 millimoles per mole [mmol/mol]) (both inclusive), as measured by central laboratory at screening
* Treatment with either:

  1. Lifestyle intervention alone
  2. 1-3 marketed oral antidiabetic drugs (OADs) (metformin, α-glucosidase inhibitors (AGI), glinides, sodium-glucose co-transporter 2 inhibitor (SGLT2i), dipeptidyl peptidase 4 (DPP4)-inhibitors, thiazolidinediones, or sulphonylureas (SU) as a single agent or in combination) according to local label
  3. Basal insulin alone or in combination with up to two marketed OADs, all according to local label

Exclusion Criteria:

* Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 60 days before screening
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Heart failure classified as being in New York Heart Association (NYHA) Class IV at screening
* Treatment with any glucagon-like peptide-1 (GLP-1) receptor agonist (RA) or a medication with GLP-1 activity within 90 days before screening
* End stage renal disease defined as estimated glomerular filtration rate (eGFR) < 15 millileters per minutes per 1.73^2 (mL/min/1.73 m^2), as measured by the central laboratory at screening
* Chronic or intermittent haemodialysis or peritoneal dialysis

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7101 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of 3-point major adverse cardiovascular event (MACE), a composite endpoint consisting of: cardiovascular (CV) death, non-fatal myocardial infarction, non-fatal stroke | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured in days.

SECONDARY OUTCOMES:
Time to first occurrence of a composite endpoint: Onset of persistent ≥40% reduction in eGFRcr (CKD-EPI), eGFRcr (CKD-EPI) <15 mL/min/1.73 m^2, Initiation of chronic kidney replacement therapy, Kidney death and CV death | From baseline (week 0) to end of study (up to 242 weeks or more)
  CKD-EPI is Chronic Kidney Disease Epidemiology Collaboration. Measured in days.
Time to first occurrence of composite endpoint consisting of: Onset of persistent macro albuminuria, ≥40% reduction in eGFRcr (CKD-EPI), eGFRcr (CKD-EPI) <15 mL/min/1.73 m^2, Initiation of chronic kidney replacement therapy and kidney death | From baseline (week 0) to end of study (up to 242 weeks or more)
  CKD-EPI is Chronic Kidney Disease Epidemiology Collaboration. Measured in days.
Time to first occurrence of an expanded 5-point MACE composite endpoint consisting of: CV death, non-fatal myocardial infarction, non-fatal stroke, coronary revascularisation and unstable angina requiring hospitalisation | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured in days.
Time to first occurrence of a composite endpoint consisting of: all-cause death, non-fatal myocardial infarction and non-fatal stroke | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured in days.
Time to first occurrence of myocardial infarction (fatal and non-fatal) | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured in days.
Time to first occurrence of stroke (fatal and non-fatal) | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured in days.
Change in eGFRcr (CKD-EPI) | From baseline (week 0) to 120 weeks
  Measured in milliliter per min per 1.73 square meter (mL/min/1.73m^2).
Ratio to baseline in Urine albumin-to-creatinine ratio (UACR) | From baseline (week 0) to 120 weeks
  Measured in ratio.
Relative change in body weight | From baseline (week 0) to 120 weeks
  Measured in percentage (%).
Change in waist circumference | From baseline (week 0) to 120 weeks
  Measured in centimeters (cm).
Change in waist-to-height ratio | From baseline (week 0) to 120 weeks
  Measured in ratio.
Change in systolic blood pressure (SBP) | From baseline (week 0) to 120 weeks
  Measured in millimeters of mercury (mmHg).
Change in diastolic blood pressure (DBP) | From baseline (week 0) to 120 weeks
  Measured in mmHg.
Ratio to baseline in lipids: Total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, very-low-density lipoprotein (VLDL) cholesterol, triglycerides and free fatty acids | From baseline (week 0) to 120 weeks
  Measured in ratio.
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to 120 weeks
  Measured in percentage-points.
Number of treatment emergent serious adverse events (TESAEs) | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured in count of events.
Number of event adjudication committee (EAC)-confirmed malignant neoplasms | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured as count of events.
Number of severe hypoglycaemic episodes (level 3) (only for participants with type 2 diabetes mellitus [T2D] at screening) | From baseline (week 0) to end of study (up to 242 weeks or more)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (617):
- United States (119):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Chambliss Clinical Trials LLC, Montgomery, Alabama
  - Honor Health, Scottsdale, Arizona
  - National Heart Institute Cal, Beverly Hills, California
  - Valley Clinical Trials, Covina, California
  - Scripps Wht Diab Inst La Jolla, La Jolla, California
  - First Valley Medical Group, Lancaster, California
  - Clinical Trials Research_Sacramento, Lincoln, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Monterey Endocrine & Diabetes Institute, Inc, Monterey, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Western University of Health Sciences, Pomona, California
  - Linda Vista Health Care Ctr, San Diego, California
  - N America Res Inst - San Dimas, San Dimas, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - Lundquist Inst.-Biom Inno-UCLA, Torrance, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Innovative Research of W FL, Clearwater, Florida
  - Florida Premier Cardiology, Delray Beach, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Life Spring Research, Miami, Florida
  - Clinical Trial Services Corp, Miami, Florida
  - Oceane 7 Medical & Research Center, Inc., Miami, Florida
  - Reyes Clinical Research, Inc, Miami, Florida
  - San Marcus Res Clin Miami Lakes, Miami Lakes, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Northeast Research Institute, Saint Augustine, Florida
  - Cardio Partners Clin Res Inst, Wellington, Florida
  - Endo Res Solutions Inc, Roswell, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Rocky Mountain Diab&Osteo Ctr, Idaho Falls, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Macoupin Research Group, Gillespie, Illinois
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - Endeavor Health, Skokie, Illinois
  - American Hlth Ntwk of IN LLC, Franklin, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Midwest Heart & Vasc Spec, Overland Park, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Louisiana Heart Center, Covington, Louisiana
  - Louisiana Heart Center, Hammond, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Clinical Trials Of America, West Monroe, Louisiana
  - Ascension Saint Agnes Heart Ca, Baltimore, Maryland
  - Elite Research Center, Flint, Michigan
  - Arcturus HC PLC Troy Med Res, Troy, Michigan
  - NDORI, Diamondhead, Mississippi
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Clinvest Research, Springfield, Missouri
  - Amicis Centers of Clinical Research, St Louis, Missouri
  - St Louis Heart & Vascular, P.C., St Louis, Missouri
  - VA Neb West Iowa Hlth System, Omaha, Nebraska
  - Methodist Physicians Clin, Omaha, Nebraska
  - Univ of NE Med Center_Omaha, Omaha, Nebraska
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Mid Hudson Med Res-New Windsor, New Windsor, New York
  - IMA Clinical Research- NY, New York, New York
  - Saratoga Clinical Research, Saratoga Springs, New York
  - Prime Global Research Inc., The Bronx, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - UNC- Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Eastern Nephr Assoc, PLLC, New Bern, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Providence Health Partners Ctr, Dayton, Ohio
  - Ohio- Advanced Medical Research, Maumee, Ohio
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Capital Area Research LLC, Newport, Pennsylvania
  - Aria Endocrine Metabolic Assoc, Philadelphia, Pennsylvania
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Baylor Scott & White Res Inst, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Dallas Heart and Vascular, Duncanville, Texas
  - Academy of Diabetes, T&E, El Paso, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - Forefront Med Res Inst PLLC, Harlingen, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Synergy Groups Medical, Houston, Texas
  - Southwest Houston Research Ltd, Houston, Texas
  - Prem Internal Med Asso Houston, Katy, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Texas Inst, Kdny & Endo Disor, Lufkin, Texas
  - Texas Institute of Cardiology PA, McKinney, Texas
  - Texas Diabetes & Endocrinology_Round Rock, Round Rock, Texas
  - Univ Of Texas Hlth Science Cntr, San Antonio, Texas
  - Clinical Advancement Ctr, PLLC, San Antonio, Texas
  - San Antonio Prem Int Med, San Antonio, Texas
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, San Antonio, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Crossroads Clinical Res- Texas, Victoria, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Valley Diab. & Endo Comp Ctr, Weslaco, Texas
  - York Clinical Research LLC, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - VA Medical Center_Salem, Salem, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Confluence Health Hospital, Wenatchee, Washington
  - Aspirus Research Institute, Wausau, Wisconsin
- Argentina (17):
  - Mautalen Salud e investigación, CABA, Buenos Aires
  - CEMEDIC, CABA, Buenos Aires
  - Hospital Italiano de la Plata, La Plata, Buenos Aires
  - Instituto Medico Catamarca, Rosario, Santa Fe Province
  - CIPREC Pueyrredon, Buenos Aires
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
  - CEDIC Centro de Investigación Clínica, CABA
  - Centro de Investigación y Prevención Cardiovascular, CABA
  - CENUDIAB Centro Médico de Nutrición v Diabetes, CABA
  - Medical Center of Diabetes and Nutrition, CABA
  - Centro de Investigaciones Metabólicas, Capital Federal
  - Instituto Médico DAMIC, Córdoba
  - Centro Médico Privado San Vicente Diabetes, Córdoba
  - Instituto de Investigaciones Clinicas, Mar del Plata
  - Consultorio Integral de Atención al Diabético, Morón
  - Instituto de Investigaciones Clinicas San Nicolás, San Nicolás
  - Sanatorio Norte, Santiago del Estero
- Australia (15):
  - Gosford Renal Research, Gosford, New South Wales
  - Paratus Clinical, Kanwal, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - GenesisCare, Auchenflower, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Royal Adelaide Hospital Cardiovascular Clinical Trials, Adelaide, South Australia
  - HeartCare SA, Leabrook, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
  - HeartCare WA (Joondalup), Joondalup, Western Australia
  - One Clinical Research, Nedlands, Western Australia
  - Clinitrials, Perth, Western Australia
- Brazil (15):
  - CPHosp Manaus Medicina, Ensino e Pesquisa LTDA, Manaus, Amazonas
  - Centro de Pesquisa em Diabetes Doenças Endócrino-Metabólicas, Fortaleza, Ceará
  - Centro de Diag. e Pesquisa da Osteoporose do Espírito Santo, Vitória, Espírito Santo
  - Núcleo de Pesquisa Clínica S/S, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - PUCCAMP - Hospital e Maternidade Celso Pierro, Campinas, São Paulo
  - i9 Pesquisas Clínicas, Campinas, São Paulo
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto, São Paulo
  - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - Instituto de Pesquisa Clinica (IPEC), São Paulo, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
  - Hospital São Lucas Copacabana, Rio de Janeiro
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
- Bulgaria (39):
  - Medical centre Asclepius OOD, Dupnitsa, Kyustendil
  - SRH - Zdrave EAD, Bankya
  - DCC - Burgas EOOD, Burgas
  - IPSOMC - Dr. Georgi Marinov, Burgas
  - Medical Centre Diamedical-2013, Dimitrovgrad
  - AIPSMC - DiMed EOOD, Haskovo
  - Medical centre Zdrave 1 OOD, Kozloduy
  - MHAT - UniHospital OOD, Panagyurishte
  - "MHAT - Pazardzhik", Pazardzhik
  - Medical center Medconsult Pleven OOD, Pleven
  - OCSOMCE - Dr. Albena Dinkova EOOD, Pleven
  - DCC Pulmed EOOD, Plovdiv
  - MHAT Med Line Clinic, Plovdiv
  - UMHAT Kaspela EOOD, Endocrinology and Metabolic Diseases Clinic, Plovdiv
  - UMHAT - Plovdiv AD, Plovdiv
  - UMHAT Pulmed, Endocrinology and Metabolic Diseases, Plovdiv
  - MHAT Sveta Karidad EAD, Plovdiv
  - MHAT Medica - Ruse OOD, Rousse
  - AIPSOMCIDEMD - Dr. Lilyana Bodurova-Troharova EOOD, Samokov
  - MHAT Dr. Ivan Seliminski - Sliven AD, Sliven
  - Nader Yabrudi - ASMPVBE Individual practice, Smolyan
  - MHAT Knyaginya Klementina - Sofia EAD, Sofia
  - MHAT Sveta Sofia EOOD, Sofia
  - Acibadem City Clinic MHAT Tokuda Department of Endocrinology and Metabolic Diseases, Sofia
  - UMHAT "Sveti Ivan Rilski" EAD, Sofia
  - UMHAT Aleksandrovska, Sofia
  - MC Orthopaedic Center Kinov EOOD, Sofia
  - Medical Institute of Ministry of interior, Sofia
  - "Medical Center Diamedical - 2013" OOD - Sofia, Sofia
  - Medical centre Vitclinic EOOD, Sofia
  - MBAL Trakia EOOD, Stara Zagora
  - Medical center Zara-Med EOOD, Stara Zagora
  - Prevencia - 2000 - MCOC OOD, Stara Zagora
  - Medical Center Nov Rehabilitatsionen center EOOD, Stara Zagora
  - UMHAT Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
  - UMHAT Sveta Marina EAD, Varna
  - DCC 1 Velingrad EOOD, Velingrad
  - Medical centre Runkovi OOD, Yambol
  - MHAT Sveti Panteleimon - Yambol AD, Yambol
- Canada (21):
  - Centricity Research Calgary, Calgary, Alberta
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Centricity Res. Barrie Endo, Barrie, Ontario
  - Centricity Research Brampton, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Clinical Research Solutions Inc., Waterloo, Ontario
  - Ctr de rech Clin de Laval, Laval, Quebec
  - Manna Research Mirabel, Mirabel, Quebec
  - Applied Medical Informatics Research, Montreal, Quebec
  - Clin des Mal Lipid de Quebec, Québec, Quebec
  - Viacar Recherche Clinique Inc., Saint-Lambert, Quebec
  - CHU-Sherbrooke, Sherbrooke, Quebec
  - Ctr de méd métab de Lanaudière, Terrebonne, Quebec
  - Recherche Clinique Sigma Inc., Québec
  - Institut universitaire de cardiologie, Québec
  - Diex Recherche Quebec Inc., Québec
- Colombia (8):
  - Servicios de Salud Ips Suramericana S.A.S., Medellín, Antioquia
  - Clinica de la Costa, Barranquilla, Atlántico
  - Fundación Hospital Universidad del Norte, Soledad, Barranquilla
  - Unidad de Estudios Clínicos de la Fundación Cardiovascular de Colombia, Bucaramanga-piedecuesta, Valle Del Menzuli - Santander, Santander Department
  - FOSCAL, Floridablanca, Santander Department
  - Fundacion del Caribe para la Investigacion Biomedica-BIOS, Barranquilla
  - CentrodeInvestigaciónenReumatologíayEspecialidadesMédicas, Bogotá
  - Somer Sociedad Medica Rionegro S.A. Somer S.A., Rionegro
- Denmark (10):
  - Herlev og Gentofte Hospital, Herlev, Capital Region
  - Aarhus Universitetshospital, Hjertesygdomme, Aarhus N, Central Jutland
  - Holbæk Sygehus, Holbæk, Region Sjælland
  - Kardiologisk Odense & Svendborg, Svendborg, Region South
  - Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus N
  - Regionshospitalet Gødstrup, Hjertesygdomme, Herning
  - Hillerød Endokrinologisk amb. H0652, Hillerød
  - Kolding Sygehus Karkirurgi, Kolding
  - Slagelse Sygehus Ambulatorium for hjertesygdomme, Slagelse
  - Viborg Sygehus, Viborg
- France (14):
  - Centre Hospitalier d'Annonay, Annonay
  - Centre Hospitalier Ardeche Nord, Annonay
  - Ap-Hp-Hopital Avicenne, Bobigny
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon-2, Grenoble
  - CH Louis Pasteur, Le Coudray
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Groupe Hospitalier Du Havre, Le Havre
  - Centre Hospitalier Universitaire de Lille-Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Montpellier-Hopital Lapeyronie, Montpellier
  - Aphp-Hopital La Pitie Salpetriere-2, Paris
  - Hopital Novo, Pontoise
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
  - RESEAU DE SANTE MUTUALISTE-Médipôle Hôpital Mutualiste, Villeurbanne
- Germany (19):
  - Diabeteszentrum-Do Dres. K U. Ch. Busch GbR, Dortmund
  - Uniklinik TU Dresden - Med. Klinik III, Dresden
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Diabetes-Zentrum Wilhelmsburg, Hamburg
  - Diabetes-Zentrum-Wilhelmsburg GbR, Hamburg
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Uniklinik Heidelberg - Innere Medizin I, Heidelberg
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Kardiologie, Leipzig
  - AmBeNet GmbH, Leipzig
  - Diabeteszentrum Ludwigsburg, Ludwigsburg
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - Uniklinik Münster, Klinik für Kardiologie I, Münster
  - Universitätsklinikum Münster - Klinik für Kardiologie I, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
  - Al-Zoebi, Wermsdorf
  - Forschungszentrum Ruhr KliFoCenter GmbH, Kahrmann, Witten
- India (74):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Lalitha Super Specialities Hospital, Guntur, Andhra Pradesh
  - Ramdev Rao Hospital, Hyderabad, Andhra Pradesh
  - Sunrise Hospital, Vijayawada, Andhra Pradesh
  - Excelcare Hospital, Guwahati, Assam
  - SMC Heart Institute and IVF Research Centre, Raipur, Chhattisgarh
  - CIMS- Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - Unicare heart institute and research centre, Surat, Gujarat
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - SSG Hospital, Baroda, Vadodara, Gujarat
  - Bankers Heart Institute, Vadodara, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - Narayana Hrudayalya Institute of Cardiac Sciences, Bangalore, Karnataka
  - Omega Hospital (P) Limited, Mangalore, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Mohak Bariatrics and Robotics, Indore, Madhya Pradesh
  - Kamalnayan Bajaj Hospital, Aurangabad, Maharashtra
  - Krishna Institute of medical sciences, Karad, Maharashtra
  - Excel Endocrine Centre, Kolhāpur, Maharashtra
  - Sir H. N. Reliance Foundation Hospital and Research Centre, Mumbai, Maharashtra
  - Wockhardt Hospital, Mumbai Central, Mumbai, Maharashtra
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - Hrudaya Cardiac and Vascular Care Centre, Nagpur, Maharashtra
  - Sengupta Hospital and Research Institute, Nagpur, Maharashtra
  - All India Institute of Medical Sciences (AIIMS), Nagpur, Nagpur, Maharashtra
  - Shalini Tai Meghe Hospital and Research Center, Nagpur, Maharashtra
  - Magnum Heart Institute, Nashik, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - Ashirwad Hospital and Research Centre, Thane, Maharashtra
  - G B Pant Institute of Postgraduate Medical Education and Research, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences_Delhi, Ansārinagar, New Delhi
  - Apollo Hospital, Delhi, New Delhi
  - AMRI Hospital, Bhubaneswar, Odisha
  - All India Institute of Medical Sciences_Khurda, Khurda, Odisha
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Fortis Heart Institute and Multispeciality Hospital, Mohali, Punjab
  - Jawahar Lal Nehru Govt. Medical College, Ajmer, Rajasthan
  - SP Medical College, Bikaner, Rajasthan
  - SMS Medical College & Attached Hospitals, Jaipur, Rajasthan
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - All India Institute of Medical Sciences (AIIMS), Jodhpur, Rajasthan
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Kg Hospital and Post Graduate Medical Institute, Coimbatore, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Guru Nanak CARE Hospitals, Hyderabad, Telangana
  - AIG Hospitals,Hyderabad, Hyderabad, Telangana
  - Diabetes Research Center, Hyderabad, Hyderabad, Telangana
  - Yashoda Hospital, Hyderabad, Telangana
  - J N Medical College, Aligarh, Uttar Pradesh
  - King George's Medical University (KGMU), Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Science, Lucknow, Uttar Pradesh
  - Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
  - IPGME&R and SSKM Hospital, Kolkata, West Bengal
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - J N Medical College, Aligarh
  - Narayana Hrudayalya Institute of Cardiac Sciences, Bangalore
  - Himachal Heart Institute, Gutkar
  - All India Institute of Medical Sciences (AIIMS), Jodhpur
  - Krishna Institute of medical sciences, Karad
  - Diabetes Care N' Research Centre Pvt. Ltd., Nagpur
  - Hrudaya Cardiac and Vascular Care Centre, Nagpur
  - Magnum Heart Institute, Nashik
  - G.B Pant Institute of Post Graduate medical education and research, New Delhi
  - BL Kapur Super Specialty Hospital, New Delhi
  - Dr. BL Kapur Memorial Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - B J Medical College & Sassoon Hospital, Pune
  - WMF's Villoo Poonawalla Memorial Hospital, Pune
  - Citi neuro centre, Telangana
- Ireland (6):
  - CRF - Galway, Galway, Connaght
  - CRF HRB - Galway, Galway, Connaght
  - Clinical Research Centre, St. Vincent's University Hospital,, Dublin, Leinster
  - Mater Miscericordiae Hospital, Dublin, Leinster
  - St James's CRF, Dublin, Leinster
  - Connolly Hospital_Blanchardstown_Diabetes Day Centre, Dublin, Leinster
- Italy (26):
  - Università degli studi G. D'Annunzio Chieti Pescara - CAST, Chieti, Abruzzo
  - A.O.U. Consorziale Policlinico di Bari, Bari, BA
  - Azienda Ospedaliero Universitaria di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliera-Universitaria Parma, Parma, Emilia-Romagna
  - Policlinico San Donato S.p.A., San Donato Milanese (MI), Lombardy
  - Ospedale Santa Maria Goretti - UOD Diabetologia, Latina, LT
  - Centro di Alta Spec. Diet., Educ. Alim. e Prev. Cardio Metab, San Donato Milanese (MI), Mi
  - ICS Maugeri, Pavia, Pv
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Rome, RM
  - AOUP Giaccone Palermo, Palermo, Sicily
  - Azienda Ospedaliera Universitaria Senese, Siena, Si
  - AOU Careggi Firenze, Florence, Tuscany
  - Azienda Ulss 3 Serenissima, Mirano, VE
  - Ente Ecclesiastico Ospedale Generale Regionale Miulli - Cardiologia e UTIC, Acquaviva delle Fonti
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - A.O.U. Bologna_ Policlinico S.Orsola Malpighi, Bologna
  - A.O.U. Policlinico S.Orsola Malpighi, Bologna
  - A.O.U policlinico "G. Rodolico-San Marco", Catania
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliero Universitaria di Modena Ospedale Civile di Baggiovara, Modena
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Pol. Uni. Campus Biomedico UOC Endocrinologia e Diabetologia, Roma
  - Pol. Uni. Campus Biomedico, Roma
  - Azienda Ospedaliero - Universitaria Sant'Andrea, Roma
  - IRCCS Multimedica, Sesto San Giovanni (MI)
- Japan (22):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Japan
  - Seino Internal Medicine Clinic, Koriyama-shi, Fukushima, Japan
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Akaicho Clinic, Chiba-shi, Chiba
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism_Diabetes Internal Medicine, Ehime
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Minami Akatsuka Clinic, Mito-shi, Ibaraki
  - Nanbu Tokushukai Hospital_Internal medicine, Okinawa
  - Osaka NISHI-UMEDA Clinic, Osaka
  - Nozaki Tokushukai Hospital_Internal medicine, Osaka
  - Yao Tokushukai General Hospital_Cardiovascular division, Osaka
  - Yao Tokushukai General Hospital, Osaka
  - Sakurabashi Watanabe Advanced Healthcare Hospital, Osaka-city, Osaka
  - Saga University Hospital, Department of Cardiology, Saga
  - Kagawa Prefectural Central Hospital, Cardiovascular Medicine, Takamatsu-shi, Kagawa
  - Takasaki General Medical Center_Department of Endocrinology / Metabolism Internal Medicine, Takasaki-shi, Gunma
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Japanese Red Cross Wakayama Medical Center_Diabetology and Endocrinology, Wakayama
  - National Hospital Organization Saitama Hospital, Wako-shi, Saitama
- Malaysia (16):
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Sultan Haji Ahmad Shah, Temerluh, Pahang
  - Hospital Seri Manjung, Seri Manjung, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Miri, Miri, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Ampang, Ampang, Selangor
  - Hospital Serdang, Kajang, Selangor
  - Hospital Melaka, Malacca
  - Hospital Putrajaya, Putrajaya
  - Hospital Miri, Sarawak
  - Hospital Ampang, Selangor Darul Ehsan
  - Hospital Shah Alam, Shah Alam
  - Hospital Putrajaya, Wilayah Persekutuan Putrajaya
- Mexico (12):
  - Centro de Investigacion Clinica Endocrinologica de Jalisco, Guadalajara, Jalisco
  - Virgen Cardiovascular Research SC, Guadalajara, Jalisco
  - Instituto de Diabetes Obesidad y Nutricion S.C., Cuernavaca, Morelos
  - Internal Medicine Clin Trials, Monterrey, Nuevo León
  - Cardiolink Clin Trials S.C., Monterrey, Nuevo León
  - Unidad Biomedica Avanzada Monterrey, Monterrey, Nuevo León
  - Clínica García Flores, Monterrey, Nuevo León
  - Centro de atención e investigación cardiovascular del Potosí, San Luis Potosí City, San Luis Potosí
  - Centro para el Desarrollo de la Medicina y la Asistencia, Culiacán, Sinaloa
  - Centro de Estudios de Investigación Metabólicos y Cardio, Ciudad Madero, Tamaulipas
  - Consultorio 1020 Hospital Angeles Xalapa, Xalapa, Veracruz
  - Promotora Medica Aguascalientes SA de CV, Aguascalientes
- Netherlands (9):
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Maxima Medisch Centrum, Eindhoven
  - Groene Hart Ziekenhuis, locatie Bleuland, Gouda
  - UMC Groningen, Groningen
  - Frisius MC Leeuwarden, Leeuwarden
  - Radboudumc, Nijmegen
  - Franciscus Gasthuis en Vlietland, Rotterdam
  - D & A Research B.V., Sneek
  - Ziekenhuis Rivierenland Tiel, Tiel
- Poland (53):
  - NSZOZ Unica CR, Dąbrówka, Greater Poland Voivodeship
  - Gierach-Med, Bygdoszcz, Kuyavian-Pomeranian Voivodeship
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów, Lesser Poland Voivodeship
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Regionalna Poradnia Diabetologiczna-Żytkiewicz-Jaruga, Stasińska Spółka Partnerska Lekarzy, Wroclaw, Lower Silesian Province
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej We Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Velocity Nova Sp. z o.o., Lublin, Lublin Voivodeship
  - ETG Poniatowa, Poniatowa, Lublin Voivodeship
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski, Lubusz Voivodeship
  - Provita Poliklinika Sp. z o.o, Warsaw, Masovian Province
  - MEDI CLINICAL Badania Kliniczne, Warsaw, Masovian Province
  - Samodzielny Publiczny Szpital Kliniczny Im. Prof. W. Orłowskiego Centrum Medycznego Kształcenia Podyplomowego, Warsaw, Masovian Voivodeship
  - ETG Warszawa Sp. z o.o., Warsaw, Masovian Voivodeship
  - Prywatna Praktyka Lekarska Anna Chudoba, Żyrardów, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku K. Kardio, Bialystok, Podlaskie Voivodeship
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok, Podlaskie Voivodeship
  - Kresmed Sp. z o. o., Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - M2M Med. Sp. z o.o. Sp. j., Chorzów, Silesian Voivodeship
  - Kardio Klinika Brynow, Katowice, Silesian Voivodeship
  - Pro Familia Altera Sp. z o.o., Katowice, Silesian Voivodeship
  - Slaskie Centrum Chorob Serca W Zabrzu, Zabrze, Silesian Voivodeship
  - Wojewodzka Poradnia dla Chorych na Cukrzyce w Zabrzu, Zabrze, Silesian Voivodeship
  - Centrum Zdrowia Metabolicznego, Poznan, Wielkopolskie Voivodeship
  - Pracownia Badan Klinicznych SALUS, Oltaszynska, Wrocław
  - Osteo-Medic s.c. A. Racewicz, J. Supronik, Bialystok
  - Renew Clinic Sp. z o.o., Bialystok
  - American Heart of Poland S.A., Bielsko-Biala
  - Centrum Medyczne Kermed Renata Bijata-Bronisz I Ewa Kowalinska Sp. j., Bydgoszcz
  - Pratia S.A., Chojnice
  - NSZOZ Unica CR, Dąbrówka
  - Centrum Kliniczno Badawcze, Elblag
  - UCK Klinika Nadcisnienia Tetniczego i Diabetologii, Gdansk
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski
  - Care Clinic Sp. z o. o., Katowice
  - Uniwersyteckie Centrum Kliniczne SUM w Katowicach, Katowice
  - Grazyna Pulka Specjalistyczny Osrodek "All-Med", Krakow
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Zanamed Medical Clinic Sp. z o.o., Lublin
  - Provita Centrum Medyczne Sp. z o.o., Piotrkow Trybunalski
  - Gaja Poradnie Lekarskie, Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej Przychodnia Specjalistyczna A Wittek H Rudzki Sp. j., Ruda Śląska
  - Polsko - Amerykanskie Kliniki Serca X Oddzial Kardiologii Inwazyjnej, Elektrofizjologii i Elektrostymulacji w Tychach, Tychy
  - Szpital Czerniakowski Sp. z o.o., Warsaw
  - BodyClinic, Warsaw
  - NASMED, Warsaw
  - Wojewodzka Poradnia dla Chorych na Cukrzyce w Zabrzu, Zabrze
  - Velocity Zamość, Zamość
  - Szpitale Powiatowe Sp. z o.o., Łask
  - American Heart of Poland S.A., Bełchatów, Łódź Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika, Lodz, Łódź Voivodeship
  - Velocity Nova Sp. z o.o., Staszów, Świętokrzyskie Voivodeship
- Isis Clinical Res. Ctr P.S.C., Guaynabo, Puerto Rico
- Serbia (9):
  - University Clinical Centre Nis, Niš, RS
  - Clinical Centre Nis, Endocrinology, Diabetes and Metabolism, Niš, RS
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocrinology department, Kragujevac
  - Policlinic for diabetes, Zaječar
- South Africa (20):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Soweto Clinical Trial Centre, Johannesburg, Gauteng
  - Hemant Makan, Johannesburg, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Ezintsha Research Centre, Johannesburg, Gauteng
  - Prinshof Medical Campus, Pretoria, Gauteng
  - Dr Seeber, Pretoria, Gauteng
  - Raslouw Private Hospital, Pretoria, Gauteng
  - Prof P. Joshi, Pretoria, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Clinical Trial Systems (CTC), Pretoria, Gauteng
  - Dr A Amod, Durban, KwaZulu-Natal
  - Netcare Umhlanga Medical Centre, Durban, KwaZulu-Natal
  - Dr Pillay's Rooms, Durban, KwaZulu-Natal
  - Lenmed Shifa Private Hospital, Durban, KwaZulu-Natal
  - Tread Research (Pty)Ltd, Cape Town, Western Cape
  - Prof Rayner_Division of Nephrology, Cape Town, Western Cape
  - Cardiac Clinical Research Unit, University of Cape Town, Cape Town, Western Cape
  - Dr Hendrik Snyman's Practice, Mossel Bay, Western Cape
  - Clinical Projects Research, Worcester, Western Cape
- Spain (18):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital de la Ribera, Alzira, Valencia
  - Hospital Comarcal de Antequera, Antequera
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Univ. de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Gregorio Marañón, Madrid
  - Hospital Clinico Virgen de la Victoria, Málaga
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Quirón, Pozuelo de Alarcón
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Virgen del Camino - Sanlúcar de Barrameda, Sanlúcar de Barrameda
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Vithas Sevilla, Seville
  - Hospital General Universitario de Toledo, Toledo
  - Hospital General de Valencia, Valencia
- Thailand (15):
  - Siriraj Hospital, Bangkok, Bangkok Noi
  - Songklanagarind Hospital, Songkhla, Had-Yai
  - Vajira Hospital - Cardio, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital_Neurology, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital_Diabetes and Endocrinology, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital_Endocrilogy, Chiang Mai
  - Rihes - Research Institute for Health Sciences, Chiang Mai
  - Chiang Rai Prachanukroh Hospital, Chiang Rai
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - Thammasat Hospital, Pathum Thani
- Turkey (Türkiye) (36):
  - Baskent University Ankara Hospital, Ankara, Bahcelievler
  - Başkent Üniversitesi Ankara Hastanesi, Ankara, Bahcelievler
  - Kartal Koşuyolu Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Istanbul, Kartal
  - Eskisehir Osmangazi University Sağlık Uygulama ve Arastirma, Eskişehir, Odunpazari
  - Eskişehir Osmangazi Üniversitesi Hastanesi- Kardiyoloji, Eskişehir, Odunpazari
  - Bursa Yüksek İhtisas Eğitim ve Araştırma Merkezi-Kardiyoloji, Bursa, Yildirim
  - T.C. Saglık Bakanlıgı Adana Sehir Egitim ve Arastirma Hastan, Adana
  - Baskent Universitesi Adana, Adana
  - Başkent Üniversitesi Adana Dr. Turgut Noyan Uygulama ve Araştırma Merkezi, Adana
  - Afyonkarahisar Health Sciences University, Afyonkarahisar
  - Afyonkarahisar Sağlık Bilimleri Üniversitesi Sağlık Uygulama Ve Araştırma Merkezi- Kardiyoloji, Afyonkarahisar
  - Ankara Bilkent Şehir Hastanesi-Dahiliye, Ankara
  - Ankara Sehir Hastanesi Dahiliye Klinigi, Ankara
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Edirne
  - Eskişehir Şehir Hastanesi- Kardiyoloji, Eskişehir
  - Istanbul University Cardiology Institute, Istanbul
  - Kanuni Sultan Suleyman Egitim ve Arastirma Hastanesi, Istanbul
  - Seyrantepe Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - Şişli Hamidiye Etfal Eğitim ve Araştırma Hastanesi- Seyrantepe Yerleşkesi- Endokrinoloji, Istanbul
  - Basaksehir Cam ve Sakura Sehir Hastanesi, Istanbul
  - Başakşehir Çam ve Sakura Şehir Hastanesi, Istanbul
  - Göztepe Prof. Dr.Süleyman Yalçın Şehir Hastanesi- Dahiliye, Istanbul
  - Dokuz Eylül Üniversitesi Araştırma Uygulama Hastanesi-Endokrinoloji, Izmir
  - Kahramanmaras Sutcu Imam University, Kahramanmaraş
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Erciyes Üniversitesi Hastanesi- Kardiyoloji, Kayseri
  - Erciyes Üniversitesi Hastanesi- Nefroloji, Kayseri
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Kocaeli Üniversitesi Hastanesi- Kardiyoloji, Kocaeli
  - Kütahya Sağlık Bilimleri Üniversitesi Evliya Çelebi EAH- Kardiyoloji, Kütahya
  - Mersin Üniversitesi Tip Fakültesi Hastanesi- Endokrinoloji, Mersin
  - Mersin University Cardiology, Mersin
  - Mersin Üniversitesi Hastanesi- Kardiyoloji, Mersin
  - Marmara Üniversitesi Pendik EAH- Endokrinoloji, Pendik/istanbul
  - Ondokuz Mayıs Üniversitesi Hastanesi- Kardiyoloji, Samsun
  - Adana Şehir Eğitim ve Araştırma Hastanesi, Yüreğir/Adana
- United Kingdom (23):
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Diabetes Centre, Heartlands Hospital, Birmingham, Birmingham, West Midlands
  - St. Richards Hospital_Cardiology, Chichester, West Sussex
  - Bradford Royal Infirmary, Bradford
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Countess of Chester Hospital - Diabetes, Chester
  - University Hospital Coventry, Coventry
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Intelligent Clinical, Glasgow
  - Hull Royal Infirmary, Hull
  - The Diabetes Centre, Ipswich
  - St James's University Hospital - Diabetes, Leeds
  - Leicester General Hospital, Leicester
  - The Good Practice, London
  - NIHR Commercial Research Delivery Centre Newcastle, Newcastle upon Tyne
  - University Dept of Medicine, Derriford Hospital, Plymouth, Plymouth
  - East Surrey Hospital, Redhill
  - Clifton Medical Centre, Rotherham
  - The Staploe Medical Centre, Soham
  - Royal Cornwall Hospital (Treliske), Truro

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com